CLINICAL TRIAL: NCT05739240
Title: Effects of Preoperative 3D Printing of Distal Intra-articular Radius Fractures on Quality of Fracture Reduction: a Randomized, Single-blinded, Monocentric Clinical Trial
Brief Title: Effects of Preoperative 3D Printing of Distal Intra-articular Radius Fractures on Quality of Fracture Reduction
Acronym: 3PAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Vilijam Zdravkovic (Other)
Responsible Party: Sponsor-Investigator, Vilijam Zdravkovic, Principal investigator, Cantonal Hospital of St. Gallen
Organization: Cantonal Hospital of St. Gallen (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22.002
Record Dates: First submitted 2023-02-12; First posted 2023-02-22 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Distal Radius Fracture; 3D Printing
MeSH Terms: conditions — Wrist Fractures | interventions — Fracture Fixation, Internal

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- no 3D model (Other)
  Interventions: Procedure: Osteosynthesis
- 3D model (Other)
  Interventions: Procedure: Osteosynthesis

INTERVENTIONS:
Procedure: Osteosynthesis — Osteosynthesis of distal radius fractures

SUMMARY:
The investigators aim to evaluate the effect of a preoperative 3D printed Model (3PAS) of distal intraarticular radius fractures on quality of fracture reduction. Surgical procedure is equal in the 3PAS and in the conventional group. To evaluate the quality of fracture reduction each patient receives a postoperative CAT-scan.

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 18 years
* Surgery criteria fulfilled
* Informed consent
* Intra-articular Fracture of the distal radius (AO 23-B and 23-C) (also including Avulsion of the processus styloideus ulnae AO/OTA 2U3A1.1) in preoperative CAT-Scan

Exclusion Criteria:

* Patient does not want a surgical treatment
* Patient does not want to participate
* Positive history for surgery due to injury of the hurt wrist beforehand
* Positive history for surgery due to injury of the opposite wrist beforehand
* Additional injuries to the hand and forearm (except distal ulna fracture AO 2U3A1.1)
* Pregnancy
* Vulnerable people
* Distal ulna fracture (except AO 2U3A1.1)
* Extraarticular radius fracture (AO 23-A)
* Concomitant injuries which interfere with the planned aftercare (intubated for a long time, additional elbow or shoulder fracture)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2024-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Articular step-off of the distal radius joint surface in the postop CAT-scan | 6 weeks
Articular gap of the distal radius joint surface in the postop CAT-scan | 6 weeks

IPD SHARING:
Plan to Share IPD: No